CLINICAL TRIAL: NCT04899063
Title: A Prospective, Multicenter Clinical Trial Designed to Evaluate the Safety and Effectiveness of the ELIOS System to Reduce Intraocular Pressure in Patients With Primary Open-Angle Glaucoma Undergoing Cataract Surgery
Brief Title: Excimer Laser Trabeculostomy Glaucoma Treatment Study
Acronym: ELTGTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elios Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP-01
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ELIOS Procedure (Other): ELIOS Procedure
  Interventions: Device: ELIOS Procedure

INTERVENTIONS:
Device: ELIOS Procedure — Treatment with the ELIOS System

SUMMARY:
Evaluation of the safety and effectiveness of the ELIOS System procedure to reduce intraocular pressure (IOP) in adult subjects with mild to moderate primary open-angle glaucoma (POAG) undergoing cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate POAG
* Operable cataract, eligible for phacoemulsification with a BCVA of 20/40 or worse
* Medicated IOP of <=24 mmHg
* Unmedicated diurnal IOP of >=22 mmHg and <=34 mmHg
* Shaffer angle grade of III or IV
* CD ratio <=0.8
* At least 45 years old

Exclusion Criteria:

* Closed-angle and secondary glaucomas
* Prior incisional glaucoma surgery, intraocular surgery, or corneal surgery
* Cannot undergo medication washout in the study eye
* Diagnosis of degenerative visual disorders
* Non-study eye with BCVA worse than 20/80
* Known corticosteroid responder
* Pregnant or nursing women; or women of childbearing potential not using medically acceptable birth control

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a decrease in medication-free mean diurnal IOP (DIOP) from baseline of at least 20% | 24 Month
  Proportion of subjects who achieve a decrease in medication-free mean diurnal IOP (DIOP) from baseline of at least 20%

SECONDARY OUTCOMES:
Mean Change in medication-free DIOP from baseline | 24 Month
  Mean change in medication-free DIOP from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal (Ike) Ahmed, MD, Study Director — Prism Eye Institute
Locations (20):
- United States (20):
  - ELIOS Vision Clinical Site, Glendale, Arizona
  - ELIOS Vision Clinical Site, Petaluma, California
  - ELIOS Vision Clinical Site, Fort Collins, Colorado
  - ELIOS Vision Clinical Site, Grand Junction, Colorado
  - ELIOS Vision Clinical Site, DeLand, Florida
  - ELIOS Vision Clinical Site, Largo, Florida
  - ELIOS Vision Clinical Site, Melbourne, Florida
  - ELIOS Vision Clinical Site, Vero Beach, Florida
  - ELIOS Vision Clinical Site, Rock Island, Illinois
  - ELIOS Vision Clinical Site, Overland Park, Kansas
  - ELIOS Vision Clinical Site, Chaska, Minnesota
  - ELIOS Vision Clinical Site, St Louis, Missouri
  - ELIOS Vision Clinical Site, Las Vegas, Nevada
  - ELIOS Vision Clinical Site, South Orange, New Jersey
  - ELIOS Vision Clinical Site, Oklahoma City, Oklahoma
  - ELIOS Vision Clinical Site, Duncanville, Texas
  - ELIOS Vision Clinical Site, El Paso, Texas
  - Elios Vision Clinical Site 2, San Antonio, Texas
  - ELIOS Vision Clinical Site, San Antonio, Texas
  - ELIOS Vision Clinical Site, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No IPD planned to be shared with other researchers